CLINICAL TRIAL: NCT07212582
Title: A Study of the Additional Human Albumin During Resuscitation in Patients With Surgical Septic Shock in Surgical Intensive Care Units: A Randomized Controlled Trial (The ALBumin Use in Surgical Septic Shock, ALBUS Study)
Brief Title: Human Albumin for Resuscitation in Surgical Septic Shock: A Randomized Controlled Trial (ALBUS Study)
Acronym: ALBUS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALBUS_SIRIRAJ
Record Dates: First submitted 2025-10-01; First posted 2025-10-08 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Critical Illness; Septic Shock
Keywords: human albumin; fluid resuscitation; colloids; Surgical Intensive Care Unit (SICU); surgical septic shock; Randomized Controlled Trial
MeSH Terms: conditions — Critical Illness; Shock, Septic | interventions — Serum Albumin, Human; Solutions; Standard of Care

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomized in a 1:1 ratio to receive either standard care alone or standard care plus intravenous 20% human albumin solution for up to 72 hours. Randomization will be performed using block randomization with a block size of 4.
Masking Description: This is an open-label study. Patients, treating clinicians, and investigators are aware of group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (Active Comparator): Patients in this group will receive standard sepsis management according to international guidelines. This includes source control, intravenous broad-spectrum antibiotics, balanced crystalloids, vasopressors, and adjunctive therapies (e.g., corticosteroids, thiamine, ventilatory and renal support) as clinically indicated. Albumin may be given if separate indications arise (e.g., perioperative use, severe hypoalbuminemia <2.5 g/dL with capillary leakage), at the discretion of the treating physician.
  Interventions: Other: Standard Care (in control arm)
- Standard Care Plus Albumin (Experimental): Patients in this group will receive standard sepsis management as above, plus intravenous 20% human albumin solution. On admission, 50 mL of 20% albumin will be infused over 2 hours, followed by additional doses for up to 72 hours, titrated according to daily serum albumin levels. The target is to maintain serum albumin >3.5 g/dL: 1 vial every 12 hours if 2.5-3.4 g/dL, or every 6 hours if <2.5 g/dL. Infusion will be withheld in the presence of fluid overload, pulmonary edema, or severe hypernatremia.
  Interventions: Drug: Human Albumin 20% Solution; Other: Standard Care (in control arm)

INTERVENTIONS:
Drug: Human Albumin 20% Solution — Intravenous 20% human albumin solution (50 mL per vial). In the experimental arm, patients receive 50 mL over 2 hours on admission, followed by additional doses for up to 72 hours, titrated to maintain serum albumin >3.5 g/dL. If albumin is 2.5-3.4 g/dL, 1 vial every 12 hours is given; if <2.5 g/dL, 1 vial every 6 hours is given. Infusion is withheld if there is fluid overload, pulmonary edema, or severe hypernatremia.
  Arms: Standard Care Plus Albumin
Other: Standard Care (in control arm) — Patients in this group will receive standard sepsis management according to international guidelines. This includes source control, intravenous broad-spectrum antibiotics, balanced crystalloids, vasopressors, and adjunctive therapies (e.g., corticosteroids, thiamine, ventilatory and renal support) as clinically indicated. Albumin may be given if separate indications arise (e.g., perioperative use, severe hypoalbuminemia <2.5 g/dL with capillary leakage), at the discretion of the treating physician.

SUMMARY:
This study will test whether giving human albumin to keep the blood albumin level above 3.5 g/dL, in addition to standard care, improves survival in patients with surgical septic shock. Septic shock is a life-threatening complication of infection that often requires urgent surgery and intensive care. Current treatment guidelines recommend intravenous fluids and medications to support blood pressure, but the best type of fluid is still uncertain.

Human albumin is a natural protein in the blood that helps maintain fluid balance and has anti-inflammatory effects. Previous studies suggest that low albumin levels are linked with worse outcomes in septic patients, and that albumin infusion might improve recovery, but results are mixed and evidence in surgical septic shock patients is lacking.

In this randomized controlled trial, adult patients with surgical septic shock admitted to the surgical intensive care unit will be randomly assigned to receive either standard care alone or standard care plus 20% human albumin solution for up to 3 days. The main outcome is survival at 28 days. Secondary outcomes include length of ICU and hospital stay, need for dialysis, ventilator-free days, vasopressor-free days, fluid balance, gastrointestinal recovery, and adverse reactions.

The results of this study will help determine whether targeted albumin replacement is beneficial in critically ill surgical patients with septic shock and could guide future fluid resuscitation strategies.

DETAILED DESCRIPTION:
This is a single-center, randomized, open-label, controlled trial designed to evaluate the effect of targeted albumin replacement in adult patients with surgical septic shock. The study will be conducted in the Surgical Intensive Care Unit at Siriraj Hospital, Bangkok, Thailand.

Eligible patients are those aged 18 years or older admitted with surgical septic shock, defined as suspected or proven surgical infection requiring an operation or surgical intervention within 48 hours, and persisting shock despite adequate initial fluid resuscitation. After informed consent, participants will be randomized in a 1:1 ratio, using block randomization, to one of two groups:

Control group: Standard sepsis management according to international guidelines, including source control, broad-spectrum antibiotics, intravenous crystalloids, vasopressors, and other adjunctive therapies as required.

Intervention group: Standard care plus intravenous 20% human albumin solution, given for up to 72 hours, with dosing guided by serum albumin levels to maintain concentrations above 3.5 g/dL.

The primary endpoint is 28-day all-cause mortality. Secondary endpoints include length of ICU and hospital stay, ventilator-free days, vasopressor-free days, 7-day cumulative fluid balance, acute kidney injury requiring renal replacement therapy, recovery of gastrointestinal function, and adverse reactions.

The planned sample size is 304 patients (152 per arm), which provides 80% power to detect a relative risk reduction of 40% in 28-day mortality (from 35% to 20%) with two-sided alpha of 0.05, accounting for 10% attrition.

Data will be analyzed primarily on an intention-to-treat basis. Interim analysis is planned after 50% enrollment to assess safety and efficacy. Both frequentist and Bayesian approaches will be applied, including logistic regression to adjust for baseline imbalances if needed.

This trial will provide evidence on whether maintaining serum albumin above 3.5 g/dL with human albumin infusion improves survival and clinical outcomes in critically ill patients with surgical septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) admitted to the surgical intensive care unit (SICU).
* Diagnosis or suspicion of surgical infection requiring surgery or surgical intervention within 48 hours of ICU admission.
* Septic shock, defined as:
* Mean arterial pressure <65 mmHg after adequate fluid resuscitation or requirement for vasopressors to maintain mean arterial pressure (MAP) ≥65 mmHg for at least 1 hour, and
* Evidence of organ dysfunction (Sequential Organ Failure Assessment (SOFA) score increase ≥2) or signs of tissue hypoperfusion (serum lactate >2 mmol/L, oliguria <0.5 mL/kg/h >2 h, or clinical evidence of poor peripheral perfusion).

Exclusion Criteria:

* Refusal of consent or do-not-resuscitate (DNR) status.
* More than 24 hours since meeting inclusion criteria.
* Contraindication to albumin infusion or history of severe allergic reaction to albumin.
* Conditions where albumin infusion is already indicated (e.g., large-volume paracentesis >5 L, hepatorenal syndrome, spontaneous bacterial peritonitis, plasmapheresis, cirrhosis, nephrotic syndrome, protein-losing enteropathy, severe burns, post-cardiac or thoracic surgery).
* Evidence of fluid overload or pulmonary edema (bilateral crepitations, chest infiltrates consistent with pulmonary edema, Central Venous Pressure >15 mmHg, Pulmonary Artery Occlusion Pressure [PAOP] >18 mmHg, or N-terminal pro-B-type Natriuretic Peptide [NT-proBNP] >900 pg/mL)
* End-stage renal disease or receiving chronic renal replacement therapy.
* Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
28-Day All-Cause Mortality | 28 days after randomization
  Mortality from any cause within 28 days of ICU admission, assessed by review of hospital records and/or telephone follow-up if the patient is discharged before Day 28.

SECONDARY OUTCOMES:
ICU Length of Stay | From ICU admission until ICU discharge or death in the ICU, assessed for up to 90 days.
  Number of days from ICU admission to ICU discharge. For participants who die in the ICU, length of stay will be recorded up to the date of death.
Hospital Length of Stay | From hospital admission until hospital discharge or in-hospital death, assessed for up to 90 days.
  Number of days from hospital admission to hospital discharge. For participants who die in the hospital, length of stay will be recorded up to the date of death.
Vasopressor-Free Days | 28 days after randomization
  Number of days alive and without vasopressor therapy during the first 28 days. Patients who die before Day 28 will be assigned zero vasopressor-free days.
7-Day Cumulative Fluid Balance | First 7 days after randomization
  Net fluid balance (total fluid input minus total output) recorded daily and summed across the first 7 days of ICU stay.
Acute Kidney Injury Requiring Renal Replacement Therapy | Up to 28 days after randomization
  Incidence of renal replacement therapy initiation for acute kidney injury, determined from ICU and hospital records.
Adverse Reactions | Up to 28 days after randomization
  Incidence of adverse reactions related to albumin infusion, including allergic or anaphylactic reactions, pulmonary edema, or electrolyte disturbances.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Siriraj Hospital, Mahidol University, Bangkok, Bangkoknoi, Thailand

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because of institutional policies at Siriraj Hospital that restrict the transfer of identifiable patient-level data outside the institution. Only aggregate, de-identified data will be reported in publications and presentations. Researchers interested in collaboration may contact the study investigators to discuss potential data analyses consistent with local regulations.